CLINICAL TRIAL: NCT06278298
Title: Different Levels of Energy of Extracorporeal Shock Wave Therapy in Post Masrectomy Lymphedema
Brief Title: Different Level of ECSWT in Post Mastectomy Lymphedema
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Christina Sabry, Senior Physical Therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/012/003318
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Lymphedema of Upper Limb
Keywords: Lymphedema, Shock wave, Breast Cancer
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Shockwave
  Interventions: Device: Shockwave
- Group B (Experimental): Shockwave
  Interventions: Device: Shockwave
- Group C (Placebo Comparator): CDT
  Interventions: Other: CDT

INTERVENTIONS:
Device: Shockwave — CDT and different dose of shockwave
  Other Names: CDT
  Arms: Group A; Group B
Other: CDT — CDT
  Arms: Group C

SUMMARY:
to investigate the effectiveness of different dosages of ECSW in the treatment of post mastectomy lymphedema volume and quality of life (Qol)

DETAILED DESCRIPTION:
The treatment program included two sessions per week for eight weeks. This study was approved by the ethical committee faculty of Physical Therapy Cairo University. All patients signed a consent form involves their agreement to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

- Criteria of selecting the patients from hospital included the following;

1. Their ages ranged from 30 to 50 years.
2. All patients were examined carefully by physician before the study procedure.
3. All patients were free from any other pathological conditions or histories of other health abnormalities except arm lymphedema.
4. They had undergone radical or modified radical mastectomy with axillary lymph node dissection with or without radiotherapy intervention.
5. Only ambulant subjects without any aides will be selected.
6. The degree of lymphedema in all subjects was grade 2 to 3 according to the classification of Foldi.(Foldi et al., 2006), (Appendix II ).
7. All patients will be medically stable.
8. Each patient will sign a consent form which in that insures her eligibility in the study.
9. All patients were treated by the same doctor and physiotherapist.

Exclusion Criteria:

* The subjects had been excluded from the study if they met one of the following criteria;

  1. The patients had recurrent malignancy, active infection, and clinical evidence of obstructive venous diseases.
  2. Patients contraindicated to ESWT due to bilateral, acute, and chronic inflammation as well as due to metastasis and poor skin condition were excluded.
  3. The patients had neurological or orthopedic problems, and diabetes.
  4. Patients with primary lymphedema.
  5. Cardiopulmonary disease which decrease the patient activites.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
lymphedema volume | two months
  tape measurment
skin thickness of the arm | two months
  ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Haytham M Elhafez, Study Director — faculty of physical therapy
Locations (1):
- Cairo University, Giza, Dokki, Egypt